CLINICAL TRIAL: NCT05929638
Title: The Effect of Aromatherapy With Lavender Essential Oil on the Sleep and Fatigue Level of Patients With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Aromatherapy With Lavender Essential Oil in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Esin Kavuran, Assist Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Esin23
Record Dates: First submitted 2023-05-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Aromatherapy; Randomized Controlled Trial; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — lavender oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Lavender oil in 15 ml opaque dark colored bottles closed with metal caps to prevent volatility to the venture group and 40 2×2 cotton pads were delivered. Patients were asked to apply lavender oil 30 minutes before going to bed. Deep breathing increases the concentration of aromatic substances in the body. The time it takes for essential oils to be absorbed into the blood circulatory system is about 30 minutes for complete absorption by the body. Information was given about dripping 3 drops of lavender oil on cotton pads and placing them 15-20 cm away from the pillow. Patients were told that they should apply lavender oil for 30 days and re-prepare the lavender oil dripped onto a new pad each night, and that the bedroom should be ventilated and free of different odors. A message was sent to the patients to remind them of the application on their phones for 30 days.
  Interventions: Behavioral: lavender oil
- Control (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Behavioral: lavender oil — The patients participating in the study were provided with the steps of applying lavender oil by inhalation, the points to be considered during the application, and the application was done in the same way by all patients.
  Arms: Experimental

SUMMARY:
The study was conducted with patients with Multiple Sclerosis (MS) who applied to the Neurology Outpatient Clinic of Atatürk University Research Hospital, met the inclusion criteria and agreed to participate in the study. At the time of the study, 96 patients were interviewed. 26 patients were excluded from the study because they did not meet the research criteria, and 70 multiple sclerosis patients constituted the research sample. 1 person from the control group and 1 person from the experimental group did not continue to work and 1 person developed a lavender allergy. The study was completed with 63 multiple sclerosis patients.

DETAILED DESCRIPTION:
Patient Description, Fatigue Severity Scale and Pittsburgh Sleep Quality Index were applied to the patients at the first interview. Lavender oil in 15 ml opaque dark colored bottles closed with metal caps to prevent volatility to the venture group (Oleum Lavandula Angustifolia/ HACCP, Halal Food, ISO 22000:2005, ISO 14001:2015, ISO 9001:2015, ISO 45001:2018) certificates) and 40 2×2 cotton pads were delivered. Studies have reported that the most common use of aromatherapy is three drops, three days a week. Patients were asked to apply lavender oil 30 minutes before going to bed. Deep breathing increases the concentration of aromatic substances in the body. The time it takes for essential oils to be absorbed into the blood circulatory system is about 30 minutes for complete absorption by the body.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Having been diagnosed with MS at least 1 year ago,
* Verbal communication (hearing and speaking)
* No problem with sense of smell,
* Not having an allergy to lavender,
* Having fatigue and sleep problems for the last 3 months,
* Not applying an intervention that helps to fall asleep,
* Pittsburgh Sleep Quality Index ≥5,
* Fatigue Severity Scale ≥4.

Exclusion Criteria:

* Having had an attack in the last month,
* Having DSM-IV Axis I disorder,
* Pregnancy,
* Using sleeping pills,
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale -FSS | two week
  The Turkish validity and reliability of the Fatigue Severity Scale, developed by Krupp et al. (1989), was determined by Armutlu et al. made by The scale is a 7-point Likert-type scale consisting of nine items. Each item is defined as 1 = strongly disagree, 7 = completely agree. The score that can be obtained from the scale varies between 9-63, and when divided by the number of items, the lowest score that can be obtained from the scale is 1 and the highest score is 7.
Pittsburgh Sleep Quality Index (PUKI) | Two week
  In 1989 Buysse et al. It was developed by Psychiatry to evaluate sleep quality in clinical studies and psychiatry practices. PSQI, which consists of 7 main headings: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleeping pills and daytime functions, evaluates sleep quality in the last month. Each subheading is evaluated between 0-3 points.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Türkoğlu, Assist.Prof., Study Chair — Ataturk University
Locations (1):
- Ataturk Unıversity, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No